CLINICAL TRIAL: NCT01436006
Title: Adult and Paediatric Patient Radiation Doses From Multidetector CT Scans: a National Survey
Brief Title: Adult and Paediatric Patient Radiation Doses From Multidetector Row Computed Tomography Scans: a National Survey
Acronym: MDCTDOSE
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Collaborators: Società Italiana di Radiologia Medica (Other)
Responsible Party: Principal Investigator, Sergio Salerno, Associate Professor, University of Palermo
Other Study IDs: MDCTDOSE/SIRM
Record Dates: First submitted 2011-07-28; First posted 2011-09-19 (Estimated); Results first posted 2015-08-04 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Cancer
Keywords: MDCT; radiation; dose
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CT scan: patient with cancer

SUMMARY:
The situation in Italy regarding radiation dose to patients undergoing Multidetector row Computed Tomography (MDCT) scans is unclear despite Italian law require that each centre check the Reference Dose Level (RDL) every two years. RDL in CT were first suggested in a document of 1998 published by the European Commission (EUR16262/1998) based on the results of an older survey in the UK from the late 1980s. Those RDLs, expressed in terms of Computed Tomography Dose Index (CTDI) and Dose Length Product (DLP), are reported in the Italian law (D.Lgs.187/00). However, in Italy there is no governmental authority comparable to the UK's National Radiological Protection Board, deputed to dose evaluation and protection.

An overview of the Italian situation is relevant in order to know the actual dose levels for MDCT administered to patients both adults and paediatrics.

DETAILED DESCRIPTION:
CT imaging is rapidly growing and now represents an indispensable medical procedure for many clinical conditions. The widespread availability and expanding use of multidetector CT (MSCT) due to its high performance and very short acquisition times, has resulted in an increase in both frequency of procedures and level of patient exposures from CT scan examinations, but issues related to radiation, including potential risks, have been relatively neglected. Particular attention should be given to CT scans in children, as they represent about 10% of all the X-ray studies performed on them, accounting for about 75% of the total dose administered. CT in children should be performed only when absolutely necessary as their longer life expectation and sensitivity to X-ray radiations may increase the risk of causing radiation-induced neoplasm's in later years.

According to the 2000 report of the United Nations Scientific Committee on the Effects of Atomic Radiation (UNSCEAR) the frequency of CT examinations in countries with high healthcare levels has increased by a factor of 8; with the mean effective dose increasing from 1,3 mSv in the 1970s to 8,8 mSv per year per 1000 persons in the early 1990s. In Switzerland, Germany and United Kingdom the increases in the number of reported CT examinations ranged between 39% and 70% over just the period 1998-2002. The 2000 ISTAT report's estimated that 1479 CT apparatus were installed in Italy performing a total of 3.327.750 CT examinations [3]. Considering an increase of 40% every 5 years, comparable to other European countries, 6.000.000 CT examinations can be estimated for 2010.

The primary objective of the study is to obtain a snapshot of Italian CT practice in adults and children that is up-to-date in regards to information concerning multidetector 16- and 64- row CT. A second goal is to update the national reference dose levels.

The study should further establish a sustainable database for the ongoing collation of further data from local surveys of CT. This will facilitate the analysis of trends and periodic review of national reference doses for CT in a way similar to other European countries.

Radiology departments dealing with adult and paediatric CT in Italy will receive an invitation to participate to the survey and a questionnaire regarding some important features of their CT equipment. Four common protocols will be used for dose calculation: CT scan of the head, lumbar spine, chest and abdomen. Cardiac CT data will be collected only for adults, as in children other examinations, such as MR are commonly preferred to CT just for radioprotection reasons.

All radiology departments using a 16 or 64 multidetector CT will be sought for enrolment in the study. Centres that perform at least 2000 MDCT examinations in either adults or paediatrics in one year and do a regular quality control on their CT scanner will be included in the survey list and divided according to their geographical site, namely the four macro-areas of Northern Italy, Centre, Southern Italy and Islands.

Each enrolled centre will receive a standardized form to fill in. The main technical parameters included in the questionnaire will be: CT scanner manufacturer, model and type, characteristics of automatic modulation system (modulation directions and chosen image quality level e.g. Noise Index and effective mAs). Tube voltage (kV), current (mA), tube rotation time(s), slice thickness, total acquisition time (s), pitch, filtration should also be given. For each patient examination Volumetric Computed Tomography Dose Index (CTDIvol) and Dose Length Product (DLP) should be collected from the dose report. For the cardiac protocol, a dedicated questionnaire will be distributed including typical cardiac parameters in addition to those mentioned above. For the protocols performed on adults, data are requested for normal patients (excluding those who were excessively small or large). For children, the age at examinations and weight are included. Paediatric studies will be those of persons less than 16 years old, as established by the Italian regulation.

In order to verify the accuracy of the console displayed values a medical physicist should measure before starting the survey the CTDIvol following the European Guidelines EUR16262/1998. Errors less then 10% between the measured and reported value will be accepted.

Each protocol will be analysed separately and descriptive statistical analysis of the main parameters will be performed. These include sample size, range, median, mean value, third quartile and percentage coefficient of variation.

The survey will be conducted over a period of twelve months. The data will be treated in an anonymous way, with the centres being coded by alphabetical letters. The investigators calculate that a sample size of 2,421 MDCT examinations for each protocol will be sufficient to guarantee a confidence of 90% and an absolute error of 5% of the average dose, with simple random sampling and assuming a conservative hypothesis that the population standard deviation is five times that estimated in a similar German survey [4].

In order to increase the accuracy of the estimation the investigators will adopt a stratified random sampling scheme that consists of stratification into the four geographical Italian macro-areas and the random selection of a number of MDCT examinations proportional to the population living in each macro-area. Stratification facilitates the tasks of data collection and survey, and aides in removing a possible source of bias related to the different frequency of MDCT apparatus, as MDCT services will be clustered into internally homogeneous strata.

ELIGIBILITY:
Inclusion Criteria:

* Patients that will be submitted to "standard" protocols for CT of the: head, chest, abdomen, lumbar spine and cardiac

Exclusion Criteria:

* Non standard MDCT examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient that will need a CT scan between March 2011 and February 2012
Sampling Method: Non-Probability Sample
Enrollment: 6700 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Salerno, Prof., Principal Investigator — University of Palermo; Daniela Origgi, PhD, Study Director — European Institute of Oncology
Locations (1):
- Azienda Ospedaliero Universitaria Policlinico, Palermo, Italy/Sicily, Italy

REFERENCES:
- [Result] Frush DP, Applegate K. Computed tomography and radiation: understanding the issues. J Am Coll Radiol. 2004 Feb;1(2):113-9. doi: 10.1016/j.jacr.2003.11.012. PMID 17411538
- [Result] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Result] Brenner DJ, Shuryak I, Einstein AJ. Impact of reduced patient life expectancy on potential cancer risks from radiologic imaging. Radiology. 2011 Oct;261(1):193-8. doi: 10.1148/radiol.11102452. Epub 2011 Jul 19. PMID 21771956

RESULTS

PARTICIPANT FLOW:
Groups:
- CT Scan: A total of 65 radiology departments, with 70 MDCT scanners, collected data of 5942 adult patients, randomly chosen, who underwent to CT examinations for common clinical for 5 common different protocols including also new examination that will be in the near future common practise as cardiac CT.
  A prevalence of multiphasic study was documented in many chest abdomen and pelvis (CAP) studies and abdominal studies.
Period: Overall Study
Arm/Group | CT Scan
Started | 6700
Completed | 6663
Not Completed | 37

BASELINE CHARACTERISTICS:
Arm/Group | CT Scan
Number analyzed (Participants) | 6700
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (16)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6080
  >=65 years | 620
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2964
  Male | 3736
Region of Enrollment [Number; unit: participants]
  Italy | 6700

OUTCOME MEASURES:

1. Primary Outcome: Value of Mean Volumetric Computed Tomography Dose Index (CTDI Vol) for Head CT Examinations.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: mGy
Groups:
- Adult: Adult patients submitted to head CT scan
- Pediatric: Pediatric patients submitted to head CT scan
Arm/Group | Adult | Pediatric
Number analyzed (Participants) | 1109 | 417
mGy | 64 (17) | 28.7 (8.2)

2. Primary Outcome: Value of Mean Volumetric Computed Tomography Dose Index (CTDI Vol) for Chest CT Examinations.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mGy
Groups:
- Chest CT- Adult: Adult patients submitted to chest CT
- Chest CT- Pediatric: Pediatric patients submitted to chest CT
Arm/Group | Chest CT- Adult | Chest CT- Pediatric
Number analyzed (Participants) | 1268 | 326
mGy | 12 (6) | 4.3 (1.7)

3. Primary Outcome: Value of Mean Volumetric Computed Tomography Dose Index (CTDI Vol) for Abdomen CT Examinations.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mGy
Groups:
- Abdomen CT Adults: Adult patients submitted to abdomen CT
- Abdomen CT Pediatric: Pediatric patients submitted to abdomen CT
Arm/Group | Abdomen CT Adults | Abdomen CT Pediatric
Number analyzed (Participants) | 1222 | 250
mGy | 15 (9) | 8.9 (3.8)

4. Primary Outcome: Value of Mean Volumetric Computed Tomography Dose Index (CTDI Vol) for Cardiac CT Examinations.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mGy
Groups:
- Adult Cardiac CT: Adult patients submitted to cardiac CT
Arm/Group | Adult Cardiac CT
Number analyzed (Participants) | 287
mGy | 43 (24)

5. Primary Outcome: Value of Mean Volumetric Computed Tomography Dose Index (CTDI Vol) for Chest Abdomen and Pelvis CT Examinations.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mGy
Groups:
- Adult Patient Chest Abdomen and Pelvis: Adult patients submitted to chest abdomen and pelvis CT examinations.
Arm/Group | Adult Patient Chest Abdomen and Pelvis
Number analyzed (Participants) | 1237
mGy | 14 (6)

6. Primary Outcome: Value of Mean Volumetric Computed Tomography Dose Index (CTDI Vol) for Spine CT Examinations.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mGy
Groups:
- CT Adult Spine: Adult patients submitted to spine CT
Arm/Group | CT Adult Spine
Number analyzed (Participants) | 584
mGy | 34 (20)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Adverse Reaction to CT: Patients submitted to CT
Arm/Group | Adverse Reaction to CT
Serious Adverse Events (participants affected / at risk) | 0/6700
Other Adverse Events (participants affected / at risk) | 0/6700

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No